CLINICAL TRIAL: NCT07284134
Title: JS107 vs Investigator's Choice as Second-line or Later Therapy for Advanced CLDN18.2-Positive Gastricor GEJ Adenocarcinoma.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS107-006-III-GC
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Injections; Irinotecan; Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): JS107: 3mg/kg, intravenous infusion, on Day 1, with a treatment cycle of every 21 days.
  Interventions: Drug: JS107 for Injection
- Control group (Active Comparator): Including 3 treatment regimens: irinotecan, paclitaxel, and docetaxel. investigators will select one regimen based on the patient's previous treatment medications, clinical benefits, and tolerability, and the administration will follow clinical guidelines and/or clinical practices. In addition, before administration, corresponding premedications (including antiemetics, preventive anti-allergy drugs, etc.) can be given with reference to clinical guidelines or drug instructions.
  Irinotecan: 150mg/m², intravenous infusion, on days 1 and 15, with a 28-day treatment cycle.
  Paclitaxel: 80mg/m², intravenous infusion, on days 1, 8, and 15, with a 28-day treatment cycle.
  Docetaxel: 75mg/m², intravenous infusion, on day 1, with a 21-day treatment cycle.
  Interventions: Drug: Irinotecan; Drug: Paclitaxel; Drug: Docetaxel

INTERVENTIONS:
Drug: JS107 for Injection — Subjects who are confirmed to meet the inclusion and exclusion criteria after screening will be randomly assigned in a 1:1 ratio to receive JS107 treatment (experimental group) or investigator's chosen treatment (control group) until the criteria for terminating the study treatment as specified in the protocol are met (including subjects experiencing BICR-confirmed radiological PD, death, loss to follow-up, withdrawal of informed consent, or termination of the study by the sponsor, whichever occurs first).
  Arms: Experimental group
Drug: Irinotecan — Subjects who are confirmed to meet the inclusion and exclusion criteria after screening will be randomly assigned in a 1:1 ratio to receive JS107 treatment (experimental group) or investigator's chosen treatment (control group) until the criteria for terminating the study treatment as specified in the protocol are met (including subjects experiencing BICR-confirmed radiological PD, death, loss to follow-up, withdrawal of informed consent, or termination of the study by the sponsor, whichever occurs first).
  Arms: Control group
Drug: Paclitaxel — Subjects who are confirmed to meet the inclusion and exclusion criteria after screening will be randomly assigned in a 1:1 ratio to receive JS107 treatment (experimental group) or investigator's chosen treatment (control group) until the criteria for terminating the study treatment as specified in the protocol are met (including subjects experiencing BICR-confirmed radiological PD, death, loss to follow-up, withdrawal of informed consent, or termination of the study by the sponsor, whichever occurs first).
  Arms: Control group
Drug: Docetaxel — Subjects who are confirmed to meet the inclusion and exclusion criteria after screening will be randomly assigned in a 1:1 ratio to receive JS107 treatment (experimental group) or investigator's chosen treatment (control group) until the criteria for terminating the study treatment as specified in the protocol are met (including subjects experiencing BICR-confirmed radiological PD, death, loss to follow-up, withdrawal of informed consent, or termination of the study by the sponsor, whichever occurs first).
  Arms: Control group

SUMMARY:
This is a multicenter, randomized, controlled, open-label, Phase III study, designed to evaluate the efficacy and safety of JS107 versus investigator-selected therapy in the second-line or later treatment of patients with advanced gastric or gastroesophageal junction adenocarcinoma positive for CLDN18.2.

The study population consists of patients with CLDN18.2-positive, HER2-negative, locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma who have received at least one prior line of systemic therapy. The primary endpoints of the study are BICR-assessed progression-free survival and overall survival.

Number of subjects and allocation:This study plans to enroll approximately 560 subjects, who will be randomized in a 1:1 ratio to receive either JS107 (experimental group) or investigator-selected therapy (control group).

DETAILED DESCRIPTION:
Patients with HER2 negative G/GEJ adenocarcinoma confirmed by histology/cytology. who have received at one prior line of systemic treatment and developed PD, and the previous treatment must include fluorouracil and platinum; CLDN18.2-positive, HER2-negative.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this study, have ICF signed after sufficient informed consent, and have good compliance.
2. Age ≥ 18 years, male or female.
3. ECOG PS 0 or 1.
4. Expected survival period≥ 3 months.
5. Patients with HER2 negative G/GEJ adenocarcinoma confirmed by histology/cytology.
6. Patients who have received at least one prior line of systemic treatments and developed PD, and the previous treatment must include fluorouracil and platinum.
7. Fresh or archival tumor tissue (blocks of formalin-fixed, paraffin-embedded [FFPE] tissue or unstained FFPE tumor tissue sections) must be available and comfirmed CLDN18.2 positivity by for central laboratory through immunohistochemistry (IHC) before randomization.
8. Having ≥ 1 measurable lesion according to RECIST v1.1 (per investigator assessment).
9. Any AEs and/or complications caused by previous therapies including surgery or radiotherapy have been adequately resolved to Grade 0 or 1 (per NCI-CTCAE v5.0 criteria) or have been stabilized in the judgment of investigators.

Exclusion Criteria:

1. Previous treatment with any drug or cellular therapy targeting CLDN18.2 (except CLDN18.2 monotarget monoclonal antibody).
2. Previously treated with an ADC loaded with a tubulin inhibitor.
3. Received strong CYP3A inhibitor or inducer within 2 weeks or 5 half-lives prior to randomization, whichever is longer.
4. Use of chemotherapy, immunotherapy or other anti-tumor therapies or participation in other clinical trials within 3 weeks prior to randomization, or use of oral fluorouracil, small molecule targeted drugs or traditional Chinese medicine for gastric cancer within 2 weeks prior to randomization.
5. Major surgery (requiring general anaesthesia and >24 hours of Hospitalisation) or other clincal trial drug treatment within 4 weeks prior to randomization, or radiotherapy within 2 weeks prior to randomization.
6. Imaging demonstrating brain metastases (except patients who have completed whole brain radiotherapy or local therapy (such as surgery), have discontinued prednisone for at least 4 weeks prior to randomization, and have stable radiologically confirmed tumor lesions and no clinical symptoms of tumor during 4 weeks prior to randomization), metastases to meninges, or spinal cord compression.
7. Tumor invades important surrounding structures (e.g., large blood vessels, trachea, etc.) with high risk of rupture and hemorrhage or airway fistula, or metastases to bone with high risk of paraplegia.
8. Thromboembolic events within 3 months prior to randomization (except patients with non-pulmonary Thromboembolism who do not require treatment or have been stably treated with anticoagulants for 14 days or longer prior to randomization).
9. History of other neoplasm malignant within 5 years prior to randomization, except for neoplasm malignant cured after treatment.
10. Having active autoimmune diseases requiring systemic treatment (i.e., immunologic modulator, corticosteroid, or Immunosuppression) within 2 years prior to randomization; replacement therapy (such as thyroid hormone, Insulin, or physiologic corticosteroid replacement therapy due to adrenal or pituitary insufficiency) is not considered systemic treatment.
11. Known severe allergic reaction to any component in the investigational drug formula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2025-12-24 (Actual); Primary Completion 2027-10-13 (Estimated); Study Completion 2028-10-17 (Estimated)

PRIMARY OUTCOMES:
BICR-PFS | up to 2 years
  Progression-Free Survival (BICR-PFS) evaluated based on Blinded Independent Central Review (BICR) (according to the RECIST v1.1 criteria)
Overall Survival | up to 5 years
  The primary endpoint of overall survival (OS) in this multicenter, randomized, open-label Phase III study is the time from randomization to death from any cause, aiming to compare the benefit between JS107 and investigator's choice of therapy in patients with CLDN18.2-positive, HER2-negative advanced gastric or gastroesophageal junction adenocarcinoma who have received at least one prior line of systemic therapy.

SECONDARY OUTCOMES:
INV-PFS | up to 2 years
  Progression-Free Survival evaluated by investigators (INV-PFS, according to the RECIST v1.1 criteria)
BICR-ORR or INV-ORR | up to 2 years
  ORR evaluated by investigators or BICR (according to the RECIST v1.1 criteria)
BICR-DCR or INV -DCR | up to 2 years
  Progression-Free Survival evaluated by investigators (INV-PFS, according to the RECIST v1.1 criteria)
BICR-DoR or INV -DoR | up to 2 years
  DoR (based on the RECIST v1.1 criteria) evaluated by investigators or BICR
The incidence rate and severity of AE | up to 2 years
  The incidence and severity of adverse events (AEs) evaluated according to the NCI-CTC AE v5.0 standard
Valley concentration of JS107 | up to 2 years
  Valley concentration of JS107 (including ADC, total antibody, and toxin)
anti-drug antibodies (ADA) for JS107 | up to 2 years
  Incidence and titer of anti-drug antibodies (ADA) for JS107 (including ADC, total antibody, and toxin)
Incidence of neutralizing antibodies (NAb) to JS107 | up to 2 years
  Incidence of neutralizing antibodies (NAb) to JS107 (including ADC, total antibody, and toxin)

OTHER OUTCOMES:
HRQOL | up to 2 years
  HRQOL (based on FACT-Ga and EORTC QLQ-C30 questionnaires)
expression levels of CLDN18.2 | up to 2 years
  Detect different expression levels of CLDN18.2 in tumor tissues and analyze the correlation with therapeutic efficacy

CONTACTS AND LOCATIONS:
Locations (68):
- China (68):
  - AnHui Provincial Cancer Hospital, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Clinical Oncology School of Fujian Medical University, Fujian Cancer Hospital, Fuzhou, Fujian
  - Union Hospital Affiliated to Fujian Medical University, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Gansu wuwei tumor hospital, Wuwei, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Nanfang hospital, Guangzhou, Guangdong
  - The sixth affiliated hospital sun yat-sen university, Guangzhou, Guangdong
  - Meizhou People's Hospital（Huangtang Hospital）, Meizhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Cancer Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Cancer Hospital Chinese Academy of Medical Sciences Langfang Campus, Langfang, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Affiliated Hospital of North China University of Technology, Tangshan, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Tumor Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Nanyang First People's Hospital National Third Class A Hospltal, Nanyang, Henan
  - Puyang People's Hospital, Puyang, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhouuniversity, Zhengzhou, Henan
  - Zhoukou Central Hospital, Zhoukou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangyang Cancer Hospital, Xiangyang, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Baotou Tumor Hospital, Baotou, Inner Mongolia
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Affiliated Hospital Of Jiangnan University, Wuxi, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Jiangxi Cancer Hospital (Jiangxi Second People's Hospital), Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Third Bethune Hospital Of Jilin University, Changchun, Jilin
  - Shengjing Hospital 0f China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital&Institute, Shenyang, Liaoning
  - General Hospital of Ningxia Medical university, Yinchuan, Ningxia
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Shandong Provincial Hospital, Ji'nan, Shandong
  - Shandong First Medical University Affiliated Tumor Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Shanghai Gobroad Cancer Hospital China Pharmaceutical University, Shanghai, Shanghai Municipality
  - The Third People's Hospital of Datong, Datong, Shanxi
  - Linfen central hospital, Linfen, Shanxi
  - First hospital of Shanxi medical university, Taiyuan, Shanxi
  - Shanxi cancer hospital, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an jiao tong University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - The second people's hospital of Yibin, Yibin, Sichuan
  - Xinjiang Medical University Affiliated Tumor Hospital, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People'S Hospital People'S Hospital of Hangzhou Medicalcollege, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No